CLINICAL TRIAL: NCT04037566
Title: A Safety Study of Autologous T Cells Engineered to Target CD19 and CRISPR Gene Edited to Eliminate Endogenous HPK1 (XYF19 CAR-T Cells) for Relapsed or Refractory Haematopoietic Malignancies.
Brief Title: CRISPR (HPK1) Edited CD19-specific CAR-T Cells (XYF19 CAR-T Cells) for CD19+ Leukemia or Lymphoma.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Xi'An Yufan Biotechnology Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Gao Guangxun, Director of Hematology Department, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V2.1
Record Dates: First submitted 2019-07-11; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Leukemia Lymphocytic Acute (ALL) in Relapse; Leukemia Lymphocytic Acute (All) Refractory; Lymphoma, B-Cell; CD19 Positive
Keywords: Leukemia Lymphocytic Acute; Lymphoma, B-Cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XYF19 CAR-T cell (Experimental): One arm study consisting of "3 + 3" dose escalation study design followed by dose expansion phase at determined MTD.
  Interventions: Genetic: XYF19 CAR-T cell; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Genetic: XYF19 CAR-T cell — Autologous T cells engineered to specify CD19 transduced with a lentiviral vector and electroporated with CRISPR guide RNA to disrupt expression of endogenous HPK1 administered by IV injection.
Drug: Cyclophosphamide — A cytotoxic chemotherapy agent used for lymphodepletion prior to XYF19 CAR-T cells.
Drug: Fludarabine — A chemotherapy agent used for lymphodepletion prior to XYF19 CAR-T cells.

SUMMARY:
This is a first-in-human trial proposed to test CD19-specific CAR-T cells with edited endogenous HPK1 (XYF19 CAR-T cells) in patients with relapsed or refractory CD19+ leukemia or lymphoma. This is an investigational study designed as a single-center, open-label and single-arm clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Subject must meet all the following criteria to be selected:

  1. Willing to provide consent/assent for participation in the study by patient or his/her legal guardian;
  2. Male or Female subjects age ≥18 and ≤55 years;
  3. Evidence of relapsed/refractory CD19+ B cell hematological malignancies. The most common relapsed/refractory B cell hematological malignancies include: (1) B cell acute lymphoblastic leukemia (B-ALL); (2) B cell lymphomas, including indolent B cell lymphoma (CLL, FL, MZL, LPL, HCL) and aggressive B cell lymphoma (DLBCL, BL, MCL)；
  4. Subjects (20 subjects of B cell acute lymphoblastic leukemia and 20 subjects of B cell lymphoma) with the following conditions:

     1. Failure to achieve complete remission (CR) after at least two lines of standard chemotherapy while not suitable for HSCT (auto/allo-HSCT)；
     2. Relapse after CR, but not eligible for HSCT (auto/allo-HSCT);
     3. Failure to achieve remission or relapse after HSCT;
  5. Leukemia patient confirmed by bone marrow aspiration that has not been alleviated; lymphoma patient with measurable or assessable lesions;
  6. Adequate organ function:

     1. Liver: ALT/AST ≥ 3 × ULN, total bilirubin ≤34.2 mol/L;
     2. Kidney: Creatinine<220 µmol/L, creatinine clearance rate (CCR) ≥ 60 mL/min;
     3. Lung: arterial oxygen saturation ≥95%;
     4. Heart: Left ventricular ejection fraction (LVEF) ≥40%;
     5. Absolute lymphocyte count (ALC) ≥ 100/μL, absolute neutrophil count (ANC) ≥ 1,000/μL, platelets (PLT) ≥ 75,000/μL;
  7. No prior anti-cancer therapy, including chemotherapy, radiotherapy, immunotherapy (immunosuppression) within 4 weeks prior to enrollment, and toxic reactions of all prior treatments recovered to grade ≤1 at the time of enrollment (except for low toxicity such as alopecia);
  8. Presence of smooth peripheral superficial venous blood flow to fulfill intravenous infusion;
  9. Karnofsky performance score ≥60; ECOG ≤2; estimated survival ≥3 months.

Exclusion Criteria:

* Subjects meeting one or more of the following criteria will be excluded:

  1. Female patient who is pregnant or breastfeeding ;
  2. Male or Female patient within Pregnancy Program in 1 year;
  3. Unwilling or unable to guarantee effective contraceptive measures (condoms or contraceptives) within 1 year after enrollment;
  4. Presence of uncontrolled infectious disease within 4 weeks prior to enrollment:
  5. Active hepatitis B or hepatitis C infection;
  6. HIV infection;
  7. Active TB;
  8. Presence of active malignancy other than disease under study, confirmed by pathology;
  9. Severe autoimmune diseases or immunodeficiency;
  10. Suffering from allergies;
  11. Joining another clinical trial within 6 weeks prior to enrollment;
  12. Using systemic corticosteroid within 4 weeks prior to enrollment (except for those who use inhaled steroids);
  13. Psychiatric disorders;
  14. History of epilepsy and seizures or other CNS pathology;
  15. Addiction to or abuse of drugs;
  16. Presence of any condition that, in the opinion of the investigator, would prohibit the patient from undergoing treatment under this protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
The adverse events associated with XYF19 CAR-T cells product will be assessed. | 30 days
  Determine safety profile of a single infusion of XYF19 CAR-T cells by monitoring the frequency and severity of adverse events assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0). Occurrence of study related adverse events defined as NCI CTCAE v5.0 > grade 3 possibly, probably, or definitely related to study treatment. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to adverse event.
Maximum tolerated dose (MTD) as determined by dose limiting toxicity (DLT). | 30 days
  The MTD is defined as the dose level at which fewer than 33% of patients experience a dose limiting toxicity (DLT). The dose limiting toxicity is defined as CTCAE grades non-reversible grade 3, or any grade 4-5 allergic reactions related to the study cell infusion; CTCAE grades non-reversible grade 3, or any grade 4-5 autoimmune reactions related to the study cell infusion; or CTCAE grades non-reversible non-hematologic grade 3, or any grade 4-5 organ toxicity (cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic) not pre-existing or due to the underlying malignancy and occurring within 30 days of study product infusion related to study cell infusion. The study will employ a standard 3+3 design to find the MTD of XYF19 CAR-T cells dose.

CONTACTS AND LOCATIONS:
Overall Officials: Guangxun GAO, Dr., Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No